CLINICAL TRIAL: NCT01785797
Title: The Effect of Subdural Drain Placement After Burr Hole Evacuation of Chronic Subdural Haematomas on Recurrence: a Prospective Randomised-controlled Multi-centre Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Peter Woo Yat Ming, Associate Consultant, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Subdural Drain Study
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Subdural Hematoma; Subdural Drain
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control: burr hole drainage only (No Intervention): Burr hole drainage of chronic subdural hematoma under general or local anesthesia without the subsequent placement of a subdural drain.
- Intervention: silicon subdural drain (Experimental): Placement of a silicon subdural drain after burr hole drainage of a chronic subdural hematoma.
  Interventions: Device: Silicon subdural drain placement after burr hole evacuation of chronic subdural hematoma

INTERVENTIONS:
Device: Silicon subdural drain placement after burr hole evacuation of chronic subdural hematoma
  Arms: Intervention: silicon subdural drain

SUMMARY:
This is a prospective randomised-controlled multi-centre trial based in Hong Kong to determine whether temporary subdural drain placement after burr hole evacuation of a chronic subdural haematoma can reduce the risk of recurrence. Consecutive patients, 60 years old or above, diagnosed to have symptomatic chronic subdural haematoma and indicated for burr hole operative drainage will be randomly allocated into one of two groups: (1) for intra-operative subdural drain placement (intervention group) or (2) not for drain placement (control group). Using web-based software block randomisation with an allocation ratio of 1:1 will be conducted. Instructions to use or not to use a drain will be contained in a sealed envelopes labelled with sequential study numbers.

Intra-operatively, if the surgeon-in-charge judges that after burr hole evacuation of the haematoma the patient's condition is unsafe for drain placement, the subject will be excluded from the study. Otherwise, randomisation will be performed at this juncture by the opening of the sealed envelop. The procedure involves placing a prefabricated silicon drain into the subdural space according to a standard protocol and will be removed on the second post-operative day at the bedside. Subjects in whom the operating surgeon judges that drain placement is unsafe will be excluded from the study. Drainage is undertaken passively by hanging the collection bag at the bedside in a dependent position. In addition to general demographic, clinical and radiological presentation data, potential risk factors for recurrence will be documented. Serial computed tomography brain scans will be arranged (before discharge, at four weeks and six months) and the occurence of significant subdural haematoma recurrence requiring repeat operative drainage at six months will be recorded. Other outcome measures to be determined at regular time intervals for a total follow-up period of six months (upon discharge, at four weeks and six months) include: functional performance in terms of the extended Glasgow Outcome Scale and modified Rankin Scale, added neurological deficit, death and other surgery-related complications. All outcomes will be documented by the trial investigators or by the responsible clinician. The data obtained will be analysed according to the principle of intention to treat.

Hypothesis: compared to burr-hole evacuation of chronic subdural haematoma alone (control), the additional placement of a subdural drain after evacuation (intervention) will reduce the risk of recurrence requiring repeat surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed to have symptomatic chronic subdural haematoma confirmed by a computed tomography or magnetic resonance imaging brain scan.
2. Ethnic Chinese
3. Age >/= 60 years-old
4. Reasonable expectation of completion of outcome measures at follow-up
5. Written informed consent

Exclusion Criteria:

1. Unsalvageable patients: fixed and dilated pupils after resuscitation or signs of brainstem herniation that precludes definitive therapy.
2. When the operating surgeon judges that drain placement may be hazardous or to be of limited benefit e.g. readily expanded brain in young patients.
3. History of previous cranial neurosurgical procedure.
4. On concurrent glucocorticoid therapy.
5. Suspected intracranial hypotension syndrome.
6. Blood dyscrasia:

   1. Use of antiplatelet medication e.g. aspirin or warfarin without adequate reversal or observation for drug effect to wear off (at least 5-7 days).
   2. Thrombocytopenia: platelet level <100 x 109/l
   3. Coagulopathy: prothrombin time PT >12sec or, activated partial thromboplastin time (APTT) >37.4 sec
7. End-stage renal/ hepatic failure.
8. Known or strong suspicion of alcohol or illicit drug abuse.
9. Pregnancy
10. Known epilepsy
11. Any neurological or non-neurological condition independent from SAH that might influence the functional outcome or other efficacy outcome measures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Significant recurrent chronic subdural hematoma i.e. requiring repeat operative drainage at six months after the primary operation | Six months after primary burr hole evacuation of chronic subdural hematoma

SECONDARY OUTCOMES:
1. Functional performance in terms of the Extended Glasgow Outcome Scale | Upon discharge, 4 weeks and 6 months after primary operation
Added neurological deficit | Upon discharge, at 4 weeks and 6 months after primary operation
Surgery-related complications | Upon discharge, at 4 weeks and 6 months after primary operation
Death | Upon discharge, at 4 weeks and 6 months after primary operation
Modified Rankin Score | Upon discharge, at 4 weeks and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China